CLINICAL TRIAL: NCT04233489
Title: Clinical Interventions to Mitigate Neurodevelopmental Risk
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The COVID-19 pandemic lead to halted protocols containing human subjects and in person interactions
Sponsor: Columbia University (Other)
Collaborators: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7857
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Child Development; Mother-Infant Interaction; Diabetes Mellitus, Gestational
Keywords: mother-infant dyad; family nurture intervention; emotional connection; synchrony; mother-infant interaction; child development; Diabetes Mellitus, Gestational
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Nurture Intervention (FNI) (Experimental): This arm contains the combined GDM+FNI and control+FNI cohort.
  Interventions: Behavioral: Family Nurture Intervention (FNI)
- Non-FNI (No Intervention): This arm contains the combined GDM+no FNI and control+no FNI cohort.

INTERVENTIONS:
Behavioral: Family Nurture Intervention (FNI) — FNI is a family based intervention that facilitates and strengthens the mother-infant emotional connection through a structured guided interaction by a physician.
  The mother is asked to sit with her baby in her arms so that they are face-to-face, and when the baby becomes restless, the physician will coach the mom to bring the baby back to a calm state. The mother will also be encouraged to verbalize her feelings to her baby. Mother-infant emotional connection is known to affect various developmental processes and improve overall health. FNI was previously shown to be efficacious in improving several long-term health outcomes in preterm infants in the neonatal intensive care unit (NICU).
  Arms: Family Nurture Intervention (FNI)

SUMMARY:
Family Nurture Intervention (FNI) has been shown to facilitate emotional connection and long-term child developmental progress in the NICU population. It has been theorized that FNI also promotes autonomic co-regulation and physiological synchrony between the mother-child dyad. The goal of the pilot study is to assess how a short one-time FNI session between at-risk mother and child dyads in the Well Baby Nursery (WBN) influences physiological synchrony, emotional connection, and developmental changes both short and long-term.

DETAILED DESCRIPTION:
The long-term objective of this work is to improve cognitive, emotional, and social developmental trajectories in at-risk children. Specially, this pilot study will assess the feasibility of Family Nurture Intervention (FNI) in the neonatal period during the infants' stay in the Well Baby Nursery (WBN) in improving developmental trajectories.

FNI is a family-based intervention that facilitates and strengthens the mother-infant emotional connection through a structured guided interaction by a trained provider. Mother-infant emotional connection is known to affect various developmental processes and improve overall health. FNI was previously shown to be efficacious in improving several long-term health outcomes in preterm infants.

In this study, the goal is to extend of the findings of FNI to another population of at risk infants - infants born to mothers suffering from gestational diabetes mellitus (GDM). These infants are generally healthy but at higher risk than controls in developing mild cognitive and motor impairments.

In this pilot phase, infants exposed to GDM and case-matched control infants will both receive FNI: (GDM+FNI and Control+FNI). These two groups will be compared to an already existing protocol and pool of participants who did not receive FNI: (GDM+no FNI and Control+no FNI). This allows the study to evaluate both GDM versus control infants as well as the presence of FNI versus no FNI.

The goal is to pilot the potential role of a short, one-time session of FNI in promoting neurodevelopment among an at-risk wellbaby nursery population. This will be achieved by comparing developmental milestones, such as cognitive and motor development, memory, attention, and emotion regulation at 6 and 15 months, between participants who received the FNI and those who did not. Another goal is to elucidate the role FNI has on autonomic co-regulation and mother-infant synchrony through physiological recordings during the FNI session in the WBN.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy mothers with and without diabetes (type 1, type 2, or gestational) and their infants
* Infants with gestational age between 37 0/7 and 40 6/7
* APGAR score above 7 five minutes after birth
* Infants between 12-72 hours of life at time of the study
* Mothers between 18-50 years old

Exclusion Criteria:

* Infants with gestational age below 37 0/7 or above 40 6/7
* Infant requiring resuscitation at birth
* Infant admitted to NICU
* Prenatal exposures to psychiatric medications, alcohol, recreational drug use, or smoking
* HIV-positive mother
* Mother with psychiatric diagnosis
* Infant with genetic disorder

Ages: 12 Hours to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Change in Welch Emotional Connection Score | Baseline and 15-months of age
  The Welch Emotional Connection Screen (WECS) is a validated scale for quantitative assessment of the emotional connection between infant and mother by scoring the interaction of the dyad in four domains: attraction, vocal communication, facial communication and sensitivity/reciprocity. Each domain is scored on a scale from 1.0 to 3.0 in 0.25 point increments, with higher scores indicating stronger emotional connection. The WECS will be measured at baseline for the FNI groups during the intervention, and at 15 months for both FNI and non-FNI groups by a researcher observing the dyadic interaction during a 3 minute period of face-to-face time. Changes in score from baseline to 15 months will be evaluated for FNI groups. Differences in emotional connection will be evaluated in FNI versus non-FNI groups by comparing WECS scores at 15-months.
Change in heart rhythm synchrony | Baseline
  Heart rhythms will be collected through non-invasive EKG monitoring of mother and infant during FNI in order to test the hypothesis that FNI improves emotional connection through autonomic synchrony. To test this, peaks will be extracted from the EKG traces of mother and infant and cross-correlation functions will be used to assess if physiological synchrony between mother-infant heart beats increases throughout the FNI session. Synchrony at the end of the session will also be used to ascertain if autonomic synchrony can be used as a predictor of WECS score or other outcomes at the follow-up sessions.
Change in Social-Emotional Questionnaire (ASQ-SE) Score | 6 months (over the phone) and 15 months (in person)
  The ASQ-SE is a 22-item parent-completed, culturally sensitive questionnaire. It is a screening tool to identify young children who may have social and emotional development trends that warrant further evaluation. It takes 10 to 15 minutes to complete. Change in score will be calculated by comparing ASQ-SE scores of FNI and non-FNI participants measuring self-regulation, compliance, communication, adaptive behaviors, autonomy, affect, and interaction with people. This would be assessed
Change in Ages and Stages questionnaire (ASQ-3) Score | 6 months (over the phone) and 15 months (in person)
  The ASQ-3 is a questionnaire aimed to pinpoint developmental progress in children between 1 month to 5.5 years in age. It is parent-centric and is administered through paper and pencil. It takes 10 to 15 minutes to complete. Change in score will be calculated by comparing ASQ-3 scores of FNI and non-FNI participants by measuring across five developmental areas: communication, gross motor, fine motor, problem solving, and personal-social.
Change in Brief Infant Toddler Social Emotional Assessment (BITSEA) score | 15 months
  BITSEA is a short 42-item parent-report screening tool used to identify social-emotional/behavioral problems and delays in competence in 12 to 36 month olds. It takes 10 to 15 minutes to complete. The measure yields two scores: a Problem Total Score and Competence Total Score. It also includes a two separate parental "worry" item for parents to rate their concern about the child's behavior and language on a 5-point scale from 1 being not at all worried to 5 being extremely worried. Change in score will be calculated by comparing BITSEA scores of FNI and non-FNI participants.

SECONDARY OUTCOMES:
Change in Parenting Stress Index (PSI-4) | 6 months (over the phone) and 15 months (in person)
  PSI-4 is a 120 item inventory designed to assess the level of stress in the parent-child relationship. It takes 5 minutes to complete. It focuses on three major domains of stress: child characteristics, parent characteristics, and situation/demographic life stress. Change in score will be calculated by comparing PSI-4 scores of mothers in FNI versus non-FNI groups. The child domain, the parent domain, and life stress domains will be compared. Child domain is separated into six subscales: distractibility, hyperactivity, adaptability, reinforces parent, demandingness, mood, and acceptability. Parent domain is separated into seven subscales: competence, isolation, attachment, health, role restriction, depression, and spouse/parenting partner relationship. Life stress provides information about factors outside the parent-child relationship.
Change in Edinburgh Postnatal Depression Scale (EPDS) | 15 months
  EPDS is a 10 question form to identify patients at risk for postnatal depression and has been proven to be an effective screening tool. Mothers who score above 13 are likely to be suffering from a depressive illness. The maximum score is 30. Those who score 10 or greater have possible depression and careful clinical assessment is suggested. The scale indicates how the mother has felt during the previous week. It takes 2 minutes to complete. Change in score will be calculated by comparing EPDS scores of mothers in FNI versus non-FNI groups.
Change in Bayley-III Scale | 15 months
  Bayley-III scale is a comprehensive tool to identify developmental delays during early childhood. It can be used between 1 and 42 months. It takes 30-45 minutes to complete. Five areas of development are assessed: cognitive, language, motor, social-emotional, and adaptive behavior. The cognitive scales comprises of 91 items to assess sensorimotor development, exploration and manipulation, object relatedness, concept formation, and memory. The language area looks at 49 items to assess receptive and 48 items to assess expressive communication. The motor domain assessed 66 items in fine motor and 71 items in gross motor. Social-emotional contains 35 items. Adaptive behavior contains 241 items. Scores for all skill areas combine to form the General Adaptive Composite (GAC) for an overall measure of development. Change in score will be calculated by comparing Bayley-III scores of FNI and non-FNI participants.
Change in Toddler Sensory Profile-2 score | 15 months
  Toddler Sensory Profile-2 evaluates a child's sensory processing patterns in the context of home, school, and community activities. Using paper and pencil or an online form, caregivers or administration fill out a questionnaire for toddlers ages 7 to 35 months. It takes 10 minutes to complete. Each form includes measurements on sensory system, behavior, sensory pattern, and school factors. Change in score will be calculated by comparing Toddler Sensory Profile-2 scores of FNI and non-FNI participants.
Change in M/CHAT R/F score | 15 months
  Modified Checklist for Autism in Toddlers, Revised, with Follow-Up (M/CHAT R/F) is a 2-stage parent-report screening tool to evaluate for Autism Spectrum Disorder (ASD) in toddlers between 16 to 30 months of age. The tool maximizes sensitivity and aims to detect as many cases of ASD as possible, and thus has high false positives. It takes 5 minutes to complete. A total score of 0-2 is low risk, 3-7 is medium, and 8-20 is high. An interview via flowchart format is also administered asking questions until a PASS or FAIL is scored. The interview is considered to screen positive if the child fails any two items on the follow-up.Change in score will be calculated by comparing M/CHAT R/F scores of FNI and non-FNI participants

CONTACTS AND LOCATIONS:
Overall Officials: Dani Dumitriu, MD/PhD, Principal Investigator — Columbia University
Locations (1):
- Morgan Stanley Children's Hospital of New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beebe B, Myers MM, Lee SH, Lange A, Ewing J, Rubinchik N, Andrews H, Austin J, Hane A, Margolis AE, Hofer M, Ludwig RJ, Welch MG. Family nurture intervention for preterm infants facilitates positive mother-infant face-to-face engagement at 4 months. Dev Psychol. 2018 Nov;54(11):2016-2031. doi: 10.1037/dev0000557. Epub 2018 Oct 4. PMID 30284883
- [Background] Isler JR, Stark RI, Grieve PG, Welch MG, Myers MM. Integrated information in the EEG of preterm infants increases with family nurture intervention, age, and conscious state. PLoS One. 2018 Oct 24;13(10):e0206237. doi: 10.1371/journal.pone.0206237. eCollection 2018. PMID 30356312
- [Background] Welch MG, Hofer MA, Brunelli SA, Stark RI, Andrews HF, Austin J, Myers MM; Family Nurture Intervention (FNI) Trial Group. Family nurture intervention (FNI): methods and treatment protocol of a randomized controlled trial in the NICU. BMC Pediatr. 2012 Feb 7;12:14. doi: 10.1186/1471-2431-12-14. Erratum In: BMC Pediatr. 2012;12:107. PMID 22314029
- [Background] Welch MG, Hofer MA, Stark RI, Andrews HF, Austin J, Glickstein SB, Ludwig RJ, Myers MM; FNI Trial Group. Randomized controlled trial of Family Nurture Intervention in the NICU: assessments of length of stay, feasibility and safety. BMC Pediatr. 2013 Sep 24;13:148. doi: 10.1186/1471-2431-13-148. PMID 24063360
- [Background] Welch MG, Firestein MR, Austin J, Hane AA, Stark RI, Hofer MA, Garland M, Glickstein SB, Brunelli SA, Ludwig RJ, Myers MM. Family Nurture Intervention in the Neonatal Intensive Care Unit improves social-relatedness, attention, and neurodevelopment of preterm infants at 18 months in a randomized controlled trial. J Child Psychol Psychiatry. 2015 Nov;56(11):1202-11. doi: 10.1111/jcpp.12405. Epub 2015 Mar 11. PMID 25763525
- [Background] Feldman R, Magori-Cohen R, Galili G, Singer M, Louzoun Y. Mother and infant coordinate heart rhythms through episodes of interaction synchrony. Infant Behav Dev. 2011 Dec;34(4):569-77. doi: 10.1016/j.infbeh.2011.06.008. Epub 2011 Jul 20. PMID 21767879